CLINICAL TRIAL: NCT05083078
Title: A Phase 1 Study to Assess the Relative PK and Tissue Distribution of Guselkumab and Risankizumab in Healthy Participants and Patients With Psoriatic Arthritis
Brief Title: A Study of Guselkumab and Risankizumab in Healthy Participants and Participants With Psoriatic Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to unanticipated feasibility constraints.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109047; 2021-000896-35 (EudraCT Number); CNTO1959PSA1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-10-11; First posted 2021-10-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Arthritis, Psoriatic; Healthy
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab; risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: Healthy Participants-Coadministration (Experimental): Healthy participants will receive a single co-administered dose of risankizumab and guselkumab subcutaneously (SC) on Day 1.
  Interventions: Drug: Guselkumab; Drug: Risankizumab
- Part 2: Psoriatic Arthritis (PsA) Participants-Coadministration (Experimental): Participants with PsA will receive a single co-administered dose of risankizumab and guselkumab SC on Day 1 and Day 29.
  Interventions: Drug: Guselkumab; Drug: Risankizumab
- Part 3: PsA Participants-Separate Administration (Experimental): Participants with PsA will receive a single dose of either risankizumab or guselkumab SC on Day 1 and Day 29.
  Interventions: Drug: Guselkumab; Drug: Risankizumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously.
  Other Names: Tremfya; CNTO1959
Drug: Risankizumab — Risankizumab will be administered subcutaneously.
  Other Names: Skyrizi

SUMMARY:
The purpose of this study is to assess the tissue distribution of guselkumab and risankizumab in healthy participants (Part 1) and psoriatic arthritis (PsA) participants (Part 2 and Part 3).

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities, must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Has a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (Coronavirus disease 2019 [COVID-19]) reverse transcription polymerase chain reaction (RT-PCR) test within 72 hours prior to study intervention administration
* Body weight within 50 kilograms (kg) to 100 kg and body mass index (BMI) within the range 18 kilograms per meter square (kg/m^2) to 30 kg/m^2 (inclusive)

Parts 2 and 3:

* Have a diagnosis of psoriatic arthritis (PsA) for at least 3 months before the first administration of study agent and meet classification criteria for psoriatic arthritis (CASPAR) at screening
* Have active plaque psoriasis

Exclusion Criteria:

Part 1:

* History or current signs and symptoms of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, genitourinary, or metabolic disturbances
* Had major illness or surgery (example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from illness or surgery, or has surgery planned during the time the participant is expected to participate in the study or within 21 weeks after the last dose of study intervention administration

Parts 2 and 3:

* History or current signs and symptoms of severe, progressive, or uncontrolled liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic (with the exception of PsA), psychiatric, genitourinary, or metabolic disturbances
* A nonplaque form of psoriasis (example, erythrodermic, guttate, or pustular)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Parts 1 , 2 and 3: Skin Tissue versus Serum Concentration Ratio | Up to Week 12
  Skin tissue versus serum concentration ratio will be summarized.
Part 1: Colon Tissue versus Serum Concentration Ratio | Up to Week 8
  Colon tissue versus serum concentration ratio will be summarized.
Parts 2 and 3: Colon Tissue versus Serum Concentration Ratio | Up to Week 4
  Colon tissue versus serum concentration ratio will be summarized.
Parts 2 and 3: Synovial Tissue versus Serum Concentration Ratio | Up to Week 12
  Synovial tissue versus serum concentration ratio will be summarized.

SECONDARY OUTCOMES:
Parts 1, 2 and 3: Maximum Observed Serum Concentration (Cmax) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  Cmax is defined as maximum observed serum concentration.
Parts 1, 2 and 3: Time to Reach Maximum Observed Serum Concentration (Tmax) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  Tmax is defined as time to reach maximum observed serum concentration.
Parts 1, 2 and 3: Area Under the Serum Concentration Versus Time Curve from Time Zero to the Time Corresponding to the Last Quantifiable Concentration (AUC[0-last]) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  AUC(0-last) is defined as area under the serum concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Parts 1, 2 and 3: Area Under the Plasma Concentration-time Curve from Time 0 to infinity (AUC[0 - Infinity]) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  AUC(0-infinity) is defined as area under the plasma concentration-time curve from time 0 to infinity with extrapolation of the terminal phase.
Parts 1, 2 and 3: Terminal Half-life (T1/2) | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  T1/2 is defined as terminal half-life.
Parts 1, 2 and 3: Apparent Total Clearance (CL/F) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  CL/F is defined as apparent total systemic clearance after extravascular administration.
Parts 1, 2 and 3: Apparent Volume of Distribution Based on Terminal Phase (Vz/F) of Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  Vz/F is defined as apparent volume of distribution based on terminal phase after extravascular administration.
Parts 1, 2 and 3: Number of Participants with Antibodies to Guselkumab and Risankizumab | Part 1: Up to Week 16, Parts 2 and 3: Up to Week 24
  The detection and characterization of antibodies to guselkumab and risankizumab will be performed using a validated assay method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency